CLINICAL TRIAL: NCT01372956
Title: Cholesterol Goal Attainment Rate and Its Associated Factors Among Dyslipidemic Patients on Lipid-lowering Drug Therapy in Korea (CRESCENDO)
Brief Title: Cholesterol Goal Attainment Rate and Its Associated Factors Among Dyslipidemic Patients on Lipid-lowering Drug Therapy in Korea
Acronym: CRESENDO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CKR-XXX-2011/1
Record Dates: First submitted 2011-06-07; First posted 2011-06-14 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Dyslipidemia
Keywords: LDL-C, cholesterol, risk factor
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dyslipidemia

SUMMARY:
This is a multi-centre, cross-sectional, chart review study to investigate cholesterol goal attainment rates defined by modified NCEP-ATP III guidelines and define its possible determinants among Korean dyslipidemic patients

DETAILED DESCRIPTION:
MC MD

ELIGIBILITY:
Inclusion Criteria:

* Patient who has a dyslipidemia with a lipid profile result within 3 months
* Patient who has a dyslipidemia without change of lipid lowering drug dosage during 3 months after lipid profile test.

Exclusion Criteria:

* Patient who involved in this study previously.
* Patient who participated in other clinical study with study drug within 90 days.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care
Sampling Method: Probability Sample
Enrollment: 4950 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Cholesterol goal attainment rate according to NCEP-ATP III guideline | Once, at enrollment

SECONDARY OUTCOMES:
Factors for cholesterol goal achievement: Age, Family history, smoking history, waist circumstance, etc. | Once, at enrollment
Cholesterol goal attainment rate related to CHD or disease history | Once, at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Ui Park, Principal Investigator — Samsung Medical Center; Jong sung Kim, Principal Investigator — Seoul National University Hospital; Sung woo Park, Principal Investigator — Kangbuk Samsung Hospital
Locations (20):
- South Korea (20):
  - Research Site, Busan, Busan
  - Research Site, Cheonan, Chungcheongnam-do
  - Research Site, Tae, Chungcheongnam-do
  - Research Site, Chuncheon, Gangwon-do
  - Research Site, Gwangju, Gwangju
  - Research Site, Anyang-si, Gyeonggi-do
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Bundang, Gyeonggi-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Guri-si, Gyeonggi-do
  - Research Site, Uijeongbu-si, Gyeonggi-do
  - Research Site, Incheon, Incheon
  - Research Site, Gwangju, Jeollabuk-do
  - Research Site, Iksan, Jeollabuk-do
  - Research Site, Daegu, Kyeongsangbuk-do
  - Research Site, Deagu, Kyeongsangbuk-do
  - Research Site, Busan, Kyeongsangnam-do
  - Research Site, Changwon, Kyeongsangnam-do
  - Research Site, Cheongju-si, North Chungcheong
  - Research Site, Seoul, Seoul